CLINICAL TRIAL: NCT04579211
Title: Prospective Analysis of Urine LAM to Eliminate NTM Sputum Screening (PAINLESS Trial)
Brief Title: Prospective Analysis of Urine LAM to Eliminate NTM Sputum Screening
Acronym: PAINLESS
Status: Enrolling by invitation | Type: Observational
Sponsor: Jerry A. Nick, M.D. (Other)
Responsible Party: Sponsor-Investigator, Jerry A. Nick, M.D., Director, Adult CF Program at National Jewish Health, National Jewish Health
Organization: National Jewish Health (Other)
Other Study IDs: NICK20A0 20-08-402-528
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with a diagnosis of CF with history of negative NTM sputum cultures: Male or female participants age 18 or greater at time of enrollment with diagnosis of CF consistent with the 2017 CFF Guidelines and NTM culture status of negative, as defined by a review of at least 3 year or more years of culture data and at least 3 NTM negative cultures with one of those negative cultures being within the last 3 years and no known history of previous positive cultures for pathogenic NTM by chart review.
  Interventions: Diagnostic Test: urine lipoarabinomannan (LAM)

INTERVENTIONS:
Diagnostic Test: urine lipoarabinomannan (LAM) — Investigate the utility of urine LAM as a test to identify individuals at very low risk for having a sputum culture positive for NTM.

SUMMARY:
This is a prospective, single-center, nonrandomized observational study to investigate the utility of urine lipoarabinomannan (LAM) as a test to identify individuals at very low risk for having a sputum culture positive for Nontuberculous Mycobacteria (NTM). The study is designed to evaluate if a urine test can eliminate the need for obtaining a sputum specimen to screen for NTM in individuals with Cystic Fibrosis (CF). The participants will be asked to provide 3 urine samples either in person or by mail over approximately 3 years. The 3 urine sample requests will be timed to coincide with their usual clinical care and routine sputum collection.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained online or in person from the participant
* Enrolled in the CFF Patient Registry (CFFPR)
* Be willing and able to adhere to study procedures in the context of clinical care, and other protocol requirements
* Diagnosis of CF consistent with the 2017 CFF Guidelines NTM culture status of negative (defined by a review of clinical and culture data with at least 3 years of clinical data available to review and at least one negative culture within the year prior to enrollment and no known history of previous positive cultures for pathogenic NTM)

Exclusion Criteria:

1. Has any other condition that, in the opinion of the Site Investigator/designee, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 adult male or female participants with a diagnosis of CF and NTM culture status of negative and no known previous positive cultures for pathogenetic NTM
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
To determine the ability of the urine LAM assay to predict continued negative sputum culture over the next 12 months. | From time enrollment to over the next 12 months
  Correlation of a negative NTM sputum culture in the year following a negative urine LAM assay

SECONDARY OUTCOMES:
To determine the ability of the urine LAM assay to predict new positive NTM sputum culture over the next 12 months. | From time of enrollment to over the next 12 months
  Correlation of a positive NTM sputum culture in the year following a positive urine LAM assay
To determine the time between a positive LAM assay and a new positive NTM culture. | 3 years
  Correlation of a positive NTM sputum culture up to 3 years following a positive urine LAM assay
To facilitate the development of a ELISA-based assay as a possible replacement to GC/MS in the clinical setting. | 3 years
  Excess urine will be used to develop and validate an alternative assay using ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A. Nick, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] De P, Amin AG, Graham B, Martiniano SL, Caceres SM, Poch KR, Jones MC, Saavedra MT, Malcolm KC, Nick JA, Chatterjee D. Urine lipoarabinomannan as a marker for low-risk of NTM infection in the CF airway. J Cyst Fibros. 2020 Sep;19(5):801-807. doi: 10.1016/j.jcf.2020.06.016. Epub 2020 Jul 3. PMID 32624408